CLINICAL TRIAL: NCT02543762
Title: Usefulness of Chromoendoscopy for the Early Detection of Colorectal Cancer Associated With Inflammatory Bowel Disease
Acronym: CE
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Complexo Hospitalario de Ourense (Other); Hospital de Manresa (Unknown); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario 12 de Octubre (Other); Hospital de Calella (Other); Hospital General de Mostoles (Other); Hospital del Mar (Other); Hospital Universitario La Fe (Other); Puerta de Hierro University Hospital (Other); Hospital Universitario de Canarias (Other); Hospital Universitari de Bellvitge (Other); Hospital de Sant Pau (Other); Complejo Hospitalario Universitario de Vigo (Other); Hospital Universitario Doctor Peset (Other)
Responsible Party: Principal Investigator, Maria Lopez Ceron, MDPHD, Hospital Clinic of Barcelona
Other Study IDs: 3-Ceron
Record Dates: First submitted 2014-05-20; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Inflammatory Bowel Disease; Colorectal Cancer
Keywords: Chromoendoscopy; Ulcerative Colitis; Crohn disease; Colorectal Neoplasia
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colorectal Neoplasms; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Inflammatory Bowel Disease: Inflammatory bowel disease (IBD) is comprised of two major disorders: ulcerative colitis and Crohn disease.
  Ulcerative colitis is a chronic inflammatory condition characterized by relapsing and remitting episodes of inflammation limited to the mucosal layer of the colon. It almost invariably involves the rectum and typically extends in a proximal and continuous fashion to involve other portions of the colon.
  Crohn disease is characterized by transmural inflammation and by skip lesions. The transmural inflammatory nature of Crohn disease may lead to fibrosis and strictures, and to obstructive clinical presentations that are not typically seen in ulcerative colitis. More commonly, the transmural inflammation results in sinus tracts, giving rise to microperforations and fistulae.
  Crohn disease may involve the entire gastrointestinal tract from mouth to perianal área patients with long-standing inflammatory bowel disease are prone to the development of colorectal cancer
  Interventions: Procedure: Chromoendoscopy

INTERVENTIONS:
Procedure: Chromoendoscopy — Chromoendoscopy involves the topical application of stains to improve tissue localization and characterization of lessions during endoscopy . Chromoendoscopy has been used in patients undergoing colonoscopy, including those undergoing surveillance for chronic ulcerative colitis. Using pit pattern classifications, chromoendoscopy has a high sensitivity and specificity for differentiating neoplastic from non-neoplastic lesions

SUMMARY:
To assess the feasibility and effectiveness of a program in L-IBD patients using CE targeted biopsies

DETAILED DESCRIPTION:
We aim to know the prevalence and incidence of dysplasia and colitis-associated colorectal cancer in patients with longstanding colonic inflammatory bowel disease (N-IBD), in Spain and the usefulness of advanced endoscopy (chromoendoscopy) for the diagnosis and endoscopic differential diagnosis of N-IBD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC or colitis EC corroborated by clinical and histology
* involvement of at least one third of the colon in patients with CD
* involvement proximal to the rectum in patients with UC
* Duration of disease > 10 years
* No clinical activity:
* May Score <6
* CDEIS <3.5

Exclusion Criteria:

* Personal history of CRC
* colectomy
* coagulopathy
* refusal to participate in the study
* known allergy to indigo carmine
* colonoscopy in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective, multicenter, multicenter study, coordinated by the Department of Gastroenterology, Hospital Clínic of Barcelona
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Prevalence and incidence of dysplasia and colitis-associated colorectal cancer in patients with longstanding colonic inflammatory bowel disease (N-IBD), in Spain | two year
  see title

SECONDARY OUTCOMES:
Usefulness of advanced endoscopy in displasia characterization (chromoendoscopy ) for the diagnosis and endoscopic differential diagnosis of NIBD. | two year
  see title

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pellise, MDPHD, Principal Investigator — Hospital Clinic of Barcelona
Locations (15):
- Spain (15):
  - Gastroenteroly Department, Hospital Clinic, Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Sant Jaume de Calella, Calella, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Manresa, Manresa, Barcelona
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Puerta del Hierro, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital general de Mostoles, Móstoles, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense, Pontevedra
  - Complexo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife
  - Hospital de la Fe, Valencia, Valencia
  - Hospital Peset, Valencia, Valencia

REFERENCES:
- [Derived] Carballal S, Maisterra S, Lopez-Serrano A, Gimeno-Garcia AZ, Vera MI, Marin-Garbriel JC, Diaz-Tasende J, Marquez L, Alvarez MA, Hernandez L, De Castro L, Gordillo J, Puig I, Vega P, Bustamante-Balen M, Acevedo J, Penas B, Lopez-Ceron M, Ricart E, Cuatrecasas M, Jimeno M, Pellise M; EndoCAR group of the Spanish Gastroenterological Association and Spanish Digestive Endoscopy Society. Real-life chromoendoscopy for neoplasia detection and characterisation in long-standing IBD. Gut. 2018 Jan;67(1):70-78. doi: 10.1136/gutjnl-2016-312332. Epub 2016 Sep 9. PMID 27612488